CLINICAL TRIAL: NCT03300011
Title: Ultrasonic Cardiogram to Evaluate the Long-term Outcome and Prognosis of Coronary Artery Chronic Total Occlusions for Percutaneous Revascularization Versus Optimal Medical Treatment
Brief Title: Ultrasonic Cardiogram Evaluate the Prognosis of Percutaneous Revascularization of Chronic Total Occlusions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Genshan Ma, Director, Southeast University, China
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 2014ZDSYLL120.1
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Coronary Chronic Total Occlusion
Keywords: ultrasonic; chronic total occlusion; heart function
MeSH Terms: interventions — Stents

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: masking for Ultrasonic Cardiogram investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- recanalisation CTO lesion successful (Experimental): Patients with CTO lesion performed PCI strategy and successfully recanalisation the CTO lesion with implanted stents .
  Interventions: Device: stent
- recanalisation CTO lesion failure (No Intervention): Patients with CTO lesion performed PCI strategy and failure recanalisation the CTO lesion with PCI wire and balloon..
- OMT (No Intervention): Patients with CTO lesion optimal medicine treatment without PCI

INTERVENTIONS:
Device: stent — PTCA or PCI
  Other Names: Balloon
  Arms: recanalisation CTO lesion successful

SUMMARY:
Chronic total occlusions (CTO) are encountered in almost one-fourth of patients undergoing coronary angiography. The presence of an untreated CTO has been related to adverse clinical prognosis, both in stable angina and acute myocardial infarction, and is often associated with persistent symptomatic angina. Depending on their symptomatic and functional status as well as anatomical complexity, CTO can be treated by optimal medical therapy only or therapy combined with coronary revascularization. This study designed to evaluate the safety and efficacy of coronary chronic total occlusion PCI by ultrasonic cardiogram.

DETAILED DESCRIPTION:
UCEPPCIOCT maintains a prospective clinical registry of all individual who undergo cardiac angiography,PCI or optimistic medicine treatment.

1. research objective to observe the changes of cardiac function postoperative PCI in patients with CTO and the incidence of major adverse cardiovascular events, and provide the reality basis for PCI strategy in clinical patients with CTO . 2. research content: follow up the patients with CTO by using echocardiography in preoperative and postoperative PCI in 1m, 3ms, 6ms, 12ms to assess the changes of cardiac structure and cardiac function. 2, comparison the 'incidence of major adverse cardiovascular events undergo PCI treatment in success and failure group in patients with CTO (such as severe angina attack, severe acute coronary syndrome, severe heart failure should be rehospitalized , fatal arrhythmia and sudden cardiac death, etc.)

ELIGIBILITY:
Inclusion Criteria:

coronary artery of chronic total occlusion

Exclusion Criteria:

ACS in 3months; once PCI or CABG; AF

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
cardiac death, | postoperation 1year
  patients with CTO postoperative sudden death cause for acute myocardial infarction or severe arrhythmia
MACE | postoperation 1year
  recurrent severe angina, revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No